CLINICAL TRIAL: NCT04316273
Title: Colonic Duplication; Two Cases Report and Review of Literature
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hamada Takrouney, clinical professor, Assiut University
Other Study IDs: IRB approval number:17300179
Record Dates: First submitted 2020-03-13; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: colonic surgery — resection of duplicated colon

SUMMARY:
Duplicated colon appendix are infrequent detected during surgical exploration. For Diagnosed cases, excision of the duplicated part is indispensable, due to risk of malignancy.

DETAILED DESCRIPTION:
Alimentary tract duplication represents(ATD) 0.2% of all pediatric congenital malformations Which affect all gastrointestinal tracts (GIT) from the mouth to the anus.

ATD more common in with no familial or racial predilection. The ileum is the most common site (30%-35%) and the colon is the least common site (7%-20%).

The transverse colon is the most common site for colonic duplication. The duplicated part of GIT maybe in the mesenteric or anti-mesenteric side. It may has same vascular supply and mesentry or not(reported only in small bowel)..

Communication between the anomalous and actual enteric lumens may or may not be present.

Here in, two cases of colonic and anal duplication add to the knowledge with review of literature of duplicated colon in children.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients till age of 18 years old
2. All patients diagnosed with duplicated colon with or without symptoms
3. Patients with duplicated colon and other associated colorectal anomalies

Exclusion Criteria:

1. Patients > 18 years with duplicated colon
2. All patients with duplication cyst

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients age group from 1 day till 18 years
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Post duplicated colon resection constipation by Bristol stool scale | 6 months
  Bristol stool form scale it range from type 1 (separate hard lumps,like hard nuts) to type 7 stool (Watery, no solid pieces ENTIRELY LIQUID)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Hamada Takrouney, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
this is case report and review of literature not more than this

REFERENCES:
- [Result] AbouZeid AA, Mohammad SA, Ibrahim SE, Fagelnor A, Zaki A. Late Diagnosis of Complete Colonic and Rectal Duplication in a Girl with an Anorectal Malformation. European J Pediatr Surg Rep. 2019 Jan;7(1):e47-e50. doi: 10.1055/s-0039-1692193. Epub 2019 Jul 5. PMID 31285983